CLINICAL TRIAL: NCT01865006
Title: Phoniatric Evaluation and Comparison of Patients Who Underwent Sutureless Thyroidectomy With Vessel Closure Devices and Conventional Total Thyroidectomy With Suture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Server Sezgin Uludag, Resident, Istanbul University
Other Study IDs: IUCTF-2013-01
Record Dates: First submitted 2013-05-21; First posted 2013-05-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Phoniatric Evaluation of Total Thyroidectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Ligasure LF1212
- Ultracision
- Conventional

SUMMARY:
The purpose of this study is to compare effect of sutureless thyroidectomy with vessel closure devices and conventional thyroidectomy with suturing on voice quality with phoniatric evaluation.

ELIGIBILITY:
Exclusion Criteria:

* Pre-operative voice problems
* Pre-operative vocal cord paralysis
* Singers and teachers
* Pre-operative known advanced stage malignity
* Previously operated for thyroid diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent to total thyroidectomy.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Voice quality change in relation with operative technique | Postoperative 1st week and 2nd month
  Voice quality change between postoperative 1st week and 2nd month in relation with operative technique (either sutureless (with Ligasure or Ultracision) or conventional technique) via Voice handicap index, videolaryngostroboscope, CSL MDVP advanced software, and Glottography.

SECONDARY OUTCOMES:
Voice quality change in relation with histopathology. | 1st week and 2nd month
  Voice quality change between postoperative 1st week and 2nd month in relation with histopathology via Voice handicap index, videolaryngostroboscope, CSL MDVP advanced software, and Glottography.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty Department of General Surgery, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Uludag SS, Teksoz S, Arikan AE, Tarhan O, Yener HM, Ozcan M, Liddy W, Randolph GW. Effect of energy-based devices on voice quality after total thyroidectomy. Eur Arch Otorhinolaryngol. 2017 May;274(5):2295-2302. doi: 10.1007/s00405-016-4444-0. Epub 2017 Feb 25. PMID 28238161